CLINICAL TRIAL: NCT00941239
Title: Gastric Tolerability and Pharmacokinetics of an Extended Release Metformin and an Immediate Release Metformin
Brief Title: Tolerability and Pharmacokinetics of Metformin and Metformin Extended Release (ER)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Laboratorios Silanes S.A. de C.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Met-LP 1007/06
Record Dates: First submitted 2009-07-15; First posted 2009-07-17 (Estimated); Last update posted 2018-01-30 (Actual); Status verified 2018-01

CONDITIONS: Healthy
Keywords: Metformin ER; Pharmacokinetics; Tolerability; Healthy volunteers
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin ER (Experimental): Extended Release Metformin
  Interventions: Drug: metformin ER
- metformin (Active Comparator): Immediate release metformin
  Interventions: Drug: metformin

INTERVENTIONS:
Drug: metformin ER — 850mg daily for 30 days
  Other Names: predial plus
  Arms: metformin ER
Drug: metformin — 850 mg daily for 30 days
  Other Names: extended release predial plus
  Arms: metformin

SUMMARY:
The purpose of this study is to determine the gastric tolerability and the pharmacokinetics of an extended release metformin compared with an immediate release metformin in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* Mexican healthy subjects with normal clinical laboratory test results and imaging (hematology, blood chemistry, urine test, VDRL, Hepatitis B, HIV, chest radiography and electrocardiogram)

Exclusion Criteria:

* Familiar or personal history of diabetes
* History of drug or alcohol abuse within the 2 years prior to the study
* A smoking habit greater than 10 cigarettes per day
* History of allergy to the study drugs
* Intercurrent disease
* Intercurrent treatment with any drug

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2007-01; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Plasmatic drug concentration | 48 hours (7.5, 15,30,45,60,75,90,120,150,180,205,240,360,480,600,720,1440,2880 min and days : 3,5,7,14,21,28,30,35)

SECONDARY OUTCOMES:
Lanza score | 30 days (0 and 30)
plasmatic glucose | 30 days (0, 6, 12 and 18 hours and days: 2,5,7,14,21,28,30 and 35)
Glycated hemoglobin | 30 days (days: 0, 14 and 30)

CONTACTS AND LOCATIONS:
Overall Officials: Oscar Torres, Ph D, Principal Investigator — UANL, Pharmacology and toxicology department; Jorge A Gonzalez, Study Director — Laboratorios Silanes S.A. de C.V.
Locations (1):
- Pharmacology and toxicology department, UANL, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Blonde L, Dailey GE, Jabbour SA, Reasner CA, Mills DJ. Gastrointestinal tolerability of extended-release metformin tablets compared to immediate-release metformin tablets: results of a retrospective cohort study. Curr Med Res Opin. 2004 Apr;20(4):565-72. doi: 10.1185/030079904125003278. PMID 15119994
- [Background] Hale TW, Kristensen JH, Hackett LP, Kohan R, Ilett KF. Transfer of metformin into human milk. Diabetologia. 2002 Nov;45(11):1509-14. doi: 10.1007/s00125-002-0939-x. Epub 2002 Sep 25. PMID 12436333
- [Background] Stumvoll M, Nurjhan N, Perriello G, Dailey G, Gerich JE. Metabolic effects of metformin in non-insulin-dependent diabetes mellitus. N Engl J Med. 1995 Aug 31;333(9):550-4. doi: 10.1056/NEJM199508313330903. PMID 7623903
- [Background] Brown BW Jr. The crossover experiment for clinical trials. Biometrics. 1980 Mar;36(1):69-79. PMID 7370374
- [Background] Schuirmann DJ. A comparison of the two one-sided tests procedure and the power approach for assessing the equivalence of average bioavailability. J Pharmacokinet Biopharm. 1987 Dec;15(6):657-80. doi: 10.1007/BF01068419. PMID 3450848
- [Background] Westlake WJ. Symmetrical confidence intervals for bioequivalence trials. Biometrics. 1976 Dec;32(4):741-4. PMID 1009222
- [Background] The United States Pharmacopeia USP26. Pags 525-526. 2003. Rockville. MD.